CLINICAL TRIAL: NCT03123705
Title: TTUHSC El Paso Public Health Biorepository (Research Core Laboratories Dental Biorepository)
Brief Title: El Paso Public Health Biorepository
Acronym: EPB
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Collaborators: The City of El Paso Department of Public Health (Unknown)
Responsible Party: Principal Investigator, Peter Rotwein, Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E16076
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Oral Disease; Bacterial Disease
MeSH Terms: conditions — Mouth Diseases; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and blood samples; bacterial and human DNA will be stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of tooth decay and other oral diseases are overlooked indicators of overall public health. To improve the understanding of oral health in El Paso, the City of El Paso Health Department will work with Texas Tech University Health Sciences Center at El Paso to determine factors that contribute to poor oral health, and lead to cavities and periodontitis. The team will collect saliva from children and young adults to study oral infections, markers of inflammation, and other contributors to oral illnesses in Mexican-American individuals.

DETAILED DESCRIPTION:
As per summary above.

ELIGIBILITY:
Inclusion Criteria:

* Individuals seen at the City of El Paso dental or pediatric clinics ages 10-21
* Healthy children and patients that are likely to be seen in the clinics within the predetermined follow-up time of 6 months

Exclusion Criteria:

* Patients under 10 years of age and over 21 years of age.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Male and female patients between the ages of 10-21.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Creation of saliva bio-repository | Through study completion, an average of 3 years
  Saliva will be collected from dental patients to be stored for research
The study of oral bacteria | Through study completion, an average of 3 years
  DNA of samples will be analyzed to determine if bacteria play a role in oral health

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Rotwein, M.D., Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information and tissue and body fluid samples will be made available to collaborating academic institutions through material transfer agreements.
Supporting Information: Study Protocol
Time Frame: Request for materials should be made after research observations are published in a peer reviewed journal.
Access Criteria: Institutions studying disease processes in Hispanic populations